CLINICAL TRIAL: NCT03378518
Title: Evaluation of Effectiveness of Blue Code Team After In-hospital Cardiopulmonary Arrest
Acronym: Codeblue
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Assistant Professor, Aydin Adnan Menderes University
Other Study IDs: Codeblue
Record Dates: First submitted 2017-12-11; First posted 2017-12-20 (Actual); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: In-hospital Cardiac Arrest
Keywords: In-hospital Cardiac Arrest, mortality

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to retrospectively examine patients evaluated by the Code Blue team on a Code Blue call in our hospital between 2016-2017.

Primary outcome: an examination of the survival rates and demographic data of the patients evaluated as an emergency by a Code Blue call in the period 2016-2017.

Secondary outcome: to determine the rates of false Code Blue calls, the clinics giving Code Blue calls and the relationship between the times of Code Blue calls and mortality.

DETAILED DESCRIPTION:
This study aimed to retrospectively examine patients evaluated by the Code Blue team on a Code Blue call in our hospital between 20016 and 2017.

Primary outcome: an examination of the survival rates and demographic data of the patients evaluated as an emergency by a Code Blue call in the period 2016-2017.Secondary outcome: to determine the rates of false Code Blue calls, the clinics giving Code Blue calls and the relationship between the times of Code Blue calls and mortality.Inclusion criteria: patients throughout the whole hospital for whom a Code Blue form was completed and who were evaluated by the Code Blue team on a Code Blue call.

ELIGIBILITY:
Inclusion criteria:

-Patients intervened by code blue team

Exclusion criteria:

* Cardiac arrest in the anesthesiology and reanimation intensive care unit
* Cardiac arrest in the newborn intensive care unit
* Out-of-hospital cardiac arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were coded blue due to in-hospital cardiac arrest between January 1, 2016 and December 31, 2016.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Blue code notification form | 12 month
  Survival rate of patients intervened by blue code team after in-hospital cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: sinan yılmaz, Principal Investigator — Aydin Adnan Menderes University
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)